CLINICAL TRIAL: NCT02601482
Title: Optimization of Interval-training in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD, PhD, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-15008542 - 2
Record Dates: First submitted 2015-11-04; First posted 2015-11-10 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glycemic control; exercise; Interval Training
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (CON) (Experimental): No exercise intervention.
  Interventions: Behavioral: CON
- Normal Interval Walking (IW-60). (Experimental): Sixty minutes with repeated cycles of 3 minutes of fast and 3 minutes of slow walking on a treadmill
  Interventions: Behavioral: IW-60
- Time-reduced Interval Walking (IW-45) (Experimental): Forty-five minutes with repeated cycles of 3 minutes of fast and 1.5 minutes of slow walking on a treadmill
  Interventions: Behavioral: IW-45

INTERVENTIONS:
Behavioral: CON
  Arms: Control (CON)
Behavioral: IW-60
  Arms: Normal Interval Walking (IW-60).
Behavioral: IW-45
  Arms: Time-reduced Interval Walking (IW-45)

SUMMARY:
A single bout of Interval-Walking (IW) exercise is superior to energy-expenditure and time-duration matched Continuous Walking (CW) exercise upon improving glycemic control. The time spend with high-intensity (fast) walking is considered to be responsible for the improvements seen, whereas the time spend with low-intensity (slow) walking is considered less important.

This study will assess if IW with maintained fast walking time duration but reduced total time duration (i.e. reduced slow walking time duration) is equally effective as IW with a normal time duration.

Subjects with type 2 diabetes will be included in a crossover, controlled study, where each subject will undergo three trials. Trials will be identical except the following interventions:

1. Sixty minutes of rest (CON)
2. Sixty minutes of classical interval walking (repeated cycles of 3 minutes of fast and 3 minutes of slow walking; IW-60)
3. Fourty-five minutes of time-reduced interval walking (repeated cycles of 3 minutes of fast and 1.5 minutes of slow walking; IW-45).

After the interventions subjects will undergo a standardized mixed meal tolerance test with assessment of glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* BMI > 25

Exclusion Criteria:

* Pregnancy
* Smoking
* Contraindication to increased levels of physical activity
* Eating disorder
* Insulin dependence

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | Within the first 4 hours after the intervention
  Glycemic control will be assessed after each intervention. Subjects will receive a standardized mixed meal tolerance test (MMTT), and blood glucose values will be obtained during the test.

SECONDARY OUTCOMES:
Matsuda insulin sensitivity index | Within the first 4 hours after the intervention
  From the measurements of glucose and insulin during the MMTT, the Matsuda index of insulin sensitivity will be assessed.
Stumvoll insulin sensitivity index | Within the first 4 hours after the intervention
  From the measurements of glucose and insulin during the MMTT, the Stumvoll index of insulin sensitivity will be assessed.
Cederholm insulin sensitivity index | Within the first 4 hours after the intervention
  From the measurements of glucose and insulin during the MMTT, the Cederholm index of insulin sensitivity will be assessed.
HOMA-2 insulin resistance index | Within the first 4 hours after the intervention
  From the measurements of glucose and insulin during the MMTT, the HOMA-2 index of insulin resistance will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Physical Activity Research (CFAS), Copenhagen, Denmark